CLINICAL TRIAL: NCT06827106
Title: Diagnostic Imaging of Temporal Bone : Technical Aspects, Applications Current and Dose-Quality Study of Differents CT Systems in Current Care
Brief Title: Dose-Quality Study in the Temporal Bone Computed Tomography in Routine Care
Status: Completed | Type: Observational
Sponsor: Aix Marseille Université (Other)
Responsible Party: Principal Investigator, IFTISSEN FRANCOIS, Médical Resident, Aix Marseille Université
Other Study IDs: Aix Marseille University
Record Dates: First submitted 2025-02-09; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Normal CT Scan; Dysplasic Disease; Tumoral Disease; Infectious Disease
Keywords: Temporal Bone; High-resolution CT scan; Spatial Resolution; Contrast-to-Noise Ratio; Radiation Dose; Diagnostic Reference Level; Observational Study; Multicenter Study; Retrospective Study; Quality Criteria; Daily Practice
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Because of the complexity of the structures studied, imaging the temporal bone requires compliance with a number of image quality criteria, in order to achieve optimum spatial resolution of the most clinically relevant anatomical landmarks. On the other hand, limiting patient exposure to ionizing radiation is a growing concern for the medical world. The challenge here is twofold: to meet a certain number of image quality criteria, in order to achieve optimum spatial resolution for the most clinically relevant anatomical landmarks, while aiming to reduce the radiation dose delivered to patients as much as possible.

Despite its routine use, few studies have compared the various commercially available solutions in terms of image quality or dose delivered, in daily practice.

The primary objective of our study is a qualitative comparison of 7 different types of CT scans on 17 anatomical structures, useful in clinical practice, taking into account the contrast-to-noise ratio (CNR).

The secondary endpoint was a comparison of radiation levels.

DETAILED DESCRIPTION:
Because of the complexity of the structures studied, imaging the temporal bone requires compliance with a number of image quality criteria, in order to achieve optimum spatial resolution of the most clinically relevant anatomical landmarks. The spatial resolution of conventional high-resolution CT is 0.5mm, whereas the dimensions of the smallest structure in the middle ear, the stapes, are of the order of 0.19mm). Despite their small size, pathological changes to these structures can have major consequences for hearing and balance, and may require exploratory or reconstructive surgery.

On the other hand, limiting patient exposure to ionizing radiation is a growing concern for the medical world, patients and public authorities alike. In the literature, effective doses vary from 50 to 970 µSv, and most protocols expose the crystalline lens (direct exposure), varying from 10 to 40 mGy in helical acquisition, depending on the technical protocol.

The International Commission on Radiological Protection has therefore proposed that the "As Low As Reasonably Achievable Radiation Exposure" (ALARA) principle should be followed, i.e. maintaining optimum spatial resolution, particularly for key anatomical landmarks in rock imaging, while reducing noise levels and radiation dose.

The challenge here is twofold: to meet a certain number of image quality criteria, in order to achieve optimum spatial resolution for the most clinically relevant anatomical landmarks, while aiming to reduce the radiation dose delivered to patients as much as possible.

Despite its routine use, few studies have compared the various commercially available solutions in terms of image quality or dose delivered, in daily practice.

To the best of our knowledge, no Diagnostic Reference Level has yet been established in the literature.

The idea would therefore be to determine objective quality criteria, based on key, clinically relevant anatomical structures, evaluated in several French centers, as part of a standard offer of care, in order to seek the right balance between the dose delivered to the patient and the quality of the image required, and thus provide clinicians with precise, reproducible tools for imaging the rock, for diagnostic or interventional purposes.

The primary objective of our study is a qualitative comparison of 7 different types of CT scans on 17 anatomical structures, useful in clinical practice, taking into account the contrast-to-noise ratio (CNR).

The secondary endpoint was a comparison of radiation levels. This is a retrospective data collection, carried out between 2023 and 2024, including 60 patients who underwent a CT scan of the temporal bone in a hospital center in mainland France, during their course of care.

Image quality was assessed independently, in a blinded fashion, by two radiologists and two ENT physicians, on the basis of a 5-point Likert semi-quantitative visual scale.

To calculate radiation exposure, the dose volume index (CTDIvol) was retrieved from the dose report for each patient, and the length-dose product (LDP) was provided automatically by the various consoles.

ELIGIBILITY:
Inclusion Criteria:

* Normal anatomy of the inner and middle ear

Exclusion Criteria:

* Motion artifacts
* Dysplastic pathologies
* Tumoral pathologies
* Infectious pathologies

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with an indication for a CT scan of the temporal bone in a hospital in mainland France
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-02-14 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
to determine temporal bone image quality criteria | 21 months
  Qualitative comparison of 17 anatomical structures according to a 5-level Likert scale

SECONDARY OUTCOMES:
to reduce the radiation dose delivered to patients | 21 months
  To compare the radiation dose received by each patient in Sievert (Sv)

CONTACTS AND LOCATIONS:
Locations (1):
- Aix Marseille University, Marseille, PACA, France

IPD SHARING:
Plan to Share IPD: No